CLINICAL TRIAL: NCT03396094
Title: Pre- and Apnoeic High Flow Oxygenation for RApid Sequence Intubation in The Emergency Department (Pre-AeRATE): a Multicentre Randomised Controlled Trial
Brief Title: Pre- and Apnoeic Oxygenation for RSI in ED
Acronym: Pre-AeRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Ng Teng Fong General Hospital (Other); Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIG17may007
Record Dates: First submitted 2018-01-01; First posted 2018-01-10 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Intubation; Oxygen Inhalation Therapy
Keywords: high flow oxygenation, rapid sequence intubation

STUDY DESIGN:
Intervention Model Description: This study consists of 2 arms (intervention and control) of parallel design. The intervention arm will receive high flow nasal cannula (HFNC) oxygenation at 60L/min for pre- and apnoeic oxygenation while the control arm will receive pre-oxygenation via non-rebreather mask and apnoeic oxygenation via nasal cannulae at 15L/min.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): High-flow nasal cannula oxygenation at 60L/min for pre-oxygenation and apnoeic oxygenation
  Interventions: Device: High-flow nasal cannulae (HFNC) oxygenation
- Control (Active Comparator): Pre-oxygenation using non-rebreather mask and apnoeic oxygenation via nasal cannulae at 15L/min
  Interventions: Device: Non-rebreather mask and standard nasal cannula

INTERVENTIONS:
Device: High-flow nasal cannulae (HFNC) oxygenation — Delivery of 60L/min of supplemental oxygen for pre-oxygenation and apnoeic oxygenation during rapid sequence intubation using the AIRVO™ 2 Humidifier with Integrated Flow Generator (Fisher & Paykel Healthcare, Auckland, New Zealand)
  Other Names: AIRVO™ 2 Humidifier with Integrated Flow Generator
  Arms: Intervention
Device: Non-rebreather mask and standard nasal cannula — Pre-oxygenation using non-rebreather mask and apnoeic oxygenation via nasal cannulae at 15L/min
  Arms: Control

SUMMARY:
Critically ill patients may need support for breathing by means of intubation, which is placement of a breathing tube into the windpipe. Rapid sequence intubation (RSI) is a method commonly used and is performed by administering medications to induce coma and muscle paralysis, followed by intubation to allow the ventilator to provide oxygen into the lungs. This procedure may be filled with potential complications.

During RSI, the patient stops spontaneous breathing after medically induced muscle paralysis occurs. Adequate oxygenation before and during paralysis is crucial to increase the reserves and prolong the time that oxygen levels in the blood remain above 90%, called the safe apnoea period. If the oxygen reserves are insufficient, the blood oxygen level will drop and can lead to permanent brain damage or even death.

This study aims to explore if delivering high-flow humidified oxygen at 60L/min via the nostrils would be superior to current methods of mask ventilation at 15L/min and nasal cannula at 15L/min, before and during paralysis respectively. If successful, this new method would allow for a longer safe apnoeic period and increase the chances for doctors to perform intubation successfully without the blood oxygen dropping below 90%.

DETAILED DESCRIPTION:
Maintaining adequate oxygenation during rapid sequence intubation (RSI) is imperative to prevent peri-intubation adverse events that can lead to increased duration of hospital and intensive care unit stay, or prolonged vegetative state requiring long-term institutionalisation.

Preliminary data from our emergency department (ED) airway registry revealed that 15% of patients experienced desaturation during intubation despite employing current best practices during RSI. In this multicentre randomised controlled trial in the ED, we aim to test the hypothesis that use of humidified high flow oxygenation via nasal cannula (HFNC) at 60L/min maintains higher oxygen saturation compared with current usual care using non-rebreather mask for preoxygenation and provides superior apnoeic oxygenation compared to the typical practice of 15L/min via standard nasal cannula.

The main goal of the study would be to improve on the lowest oxygen saturation during intubation, and thereby increase the safe apnoeic time during RSI. We plan to enrol adult patients who require rapid sequence intubation due to medical, surgical or traumatic conditions in the EDs of National University Hospital and Ng Teng Fong General Hospital.

Eligible patients will undergo block randomisation at equal ratio into 2 possible treatment combinations of pre-oxygenation and apnoeic oxygenation. The primary endpoint will be the lowest oxygen saturation achieved from time of administration of paralytic agent until quantitative end-tidal carbon dioxide is detected for the first intubation attempt.

Higher failure rates for intubation in unfasted patients in the ED compared to fasted patients in elective settings increase the risk of aspiration if re-oxygenation is required with bag-valve-mask ventilation. Prolongation of safe apnoea time through maintenance of oxygen saturation above 90% using HFNC oxygenation during RSI could potentially change current clinical practice, improve standard of care and translate to better outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 21 years and above, who require RSI due to medical, surgical and traumatic conditions, in the Emergency Departments of NUH and Ng Teng Fong General Hospital (NTFGH)

Exclusion Criteria:

* Patients with "do-not-resuscitate" orders
* Crash, awake or delayed sequence intubations
* Patients requiring non-invasive positive pressure ventilation
* Cardiac arrest
* Clinical suspicion or confirmed diagnosis of base of skull fractures or severe facial trauma that precludes nasal cannula placement
* Vulnerable patient populations (e.g. pregnant women, prisoners)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Lowest SpO2 achieved during first intubation attempt | From time of administration of paralytic agent until quantitative ETCO2 is detected post-intubation up to 45 minutes
  Lowest SpO2 achieved during first intubation attempt which is defined as first attempt to insert endotracheal tube into oropharynx

SECONDARY OUTCOMES:
Number of attempts at intubation | Number of attempts required until successful intubation up to 45 minutes or termination of procedure, whichever is earlier
  Number of attempts until successful intubation as indicated by detection of quantitative ETCO2
Safe apnoea time during intubation | From start of paralysis to time when SpO2 drops to less than 90% up to 45 minutes
  Duration of apnoea where SpO2 remains ≥ 90%
Incidence of SpO2 < 90% | From start of paralysis to successful intubation up to 45 minutes
  Incidence of SpO2 < 90% during apnoea
Peri-intubation adverse events | From induction to 15 minutes after intubation
  Peri-intubation adverse events defined as hypotension, hypertension, tachycardia, bradycardia, regurgitation, aspiration, cardiac arrhythmia, cardiac arrest during RSI, oropharynx or dental trauma
Length of time to successful intubation | From induction until successful intubation as confirmed by detection of quantitative ETCO2 up to 45 minutes
  Time taken from induction to successful intubation attempt

CONTACTS AND LOCATIONS:
Overall Officials: Mui Teng Chua, MBBS, MPH, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chua MT, Khan FA, Ng WM, Lu Q, Low MJW, Yau YW, Punyadasa A, Kuan WS. Pre- and Apnoeic high flow oxygenation for RApid sequence intubation in The Emergency department (Pre-AeRATE): study protocol for a multicentre, randomised controlled trial. Trials. 2019 Apr 4;20(1):195. doi: 10.1186/s13063-019-3305-8. PMID 30947740

DOCUMENTS (1):
  • Study Protocol (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/94/NCT03396094/Prot_000.pdf